CLINICAL TRIAL: NCT00872573
Title: Prospective, Uncontrolled, Two-centre, RSA, Post-market Surveillance Study to Evaluate the Stability of the C-Stem™ AMT Femoral Component in Primary Total Hip Arthroplasty.
Brief Title: A Two Centre Study to Assess the Stability and Long-term Performance of the C-Stem™ AMT in a Total Primary Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Technical issues with RSA at main site and departure of Principal Investigator
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT03/14
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cemented
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-Stem™ AMT Femoral Component (Other)
  Interventions: Device: C-Stem™ AMT Femoral Component (standard and high off-set variants)

INTERVENTIONS:
Device: C-Stem™ AMT Femoral Component (standard and high off-set variants) — A polished triple tapered cemented femoral component for use in total hip replacement

SUMMARY:
The purpose of this study is to monitor the stability of the C-Stem™ AMT hip within the thigh bone when used in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be evaluated at regular intervals following hip surgery using patient, clinical, standard x-ray assessments and special x-rays which allow the stability of the implant to be determined.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 60 and 80 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects undergoing primary total hip replacement that are considered suitable for a cemented femoral stem and metal femoral head and an all polyethylene acetabular cup.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Subjects undergoing revision hip replacement

iii) Subjects undergoing simultaneous bilateral hip replacements.

iv) Subjects with a contralateral hip replacement, which was implanted less than six months previously or is not performing satisfactorily.

v) Women who are pregnant.

vi) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

vii) Subjects who have participated in a clinical study with an investigational product in the last 12 months.

viii) Subjects who are currently involved in any injury litigation claims.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-01 (Actual)

PRIMARY OUTCOMES:
Distal migration of the femoral stem at the 5-year time point | 5 years

SECONDARY OUTCOMES:
ML/AP translation and all rotations out to 5 years | pre-discharge, 3mths, 6mths, 1yr, 18mths, 2yrs, 3yrs and 5yrs post-surgery
Harris Hip score | 3mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery
Oxford Hip score | 3mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery
Radiological analysis | 3mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- North Bristol NHS Trust, Bristol, United Kingdom